CLINICAL TRIAL: NCT00180219
Title: An Open Clinical Trial to Assess the Influence of Gestational Stage and Maternal Age on Arterial Stiffness of the Mother (Hormonal and Age Related Changes of the Aortal Elasticity)
Brief Title: Clinical Trial to Assess the Influence of Gestational Stage and Maternal Age on Arterial Stiffness of the Mother
Status: Withdrawn | Type: Observational
Why Stopped: recruitment failure
Sponsor: Technische Universität Dresden (Other)
Other Study IDs: IKPD-S-01-04
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy Trimester, First; Pregnancy Trimester, Second; Pregnancy Trimester, Third
Keywords: G08.520.769.550.408; G08.520.769.550.490; G08.520.769.550.520
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 20 to 22 years
- 2: 30 to 32 years
- 3: 40 to 42 years

SUMMARY:
This is a single-centre, open, parallel-group study with three age groups; no study medication or intervention will be provided. This is a longitudinal follow-up of physiological parameters.

DETAILED DESCRIPTION:
The subjects will be investigated as outpatients. For each subject, 4 individual dates with a duration of approximately 30 minutes each are scheduled - at the end of the first trimenon, at the end of the second trimenon, 4 weeks prior to the calculated date of birth, and 6 weeks after the effective date of birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women without major concomitant disease
* Willing and able to provide informed consent
* Age (three age groups):

  * 20 to 22 years
  * 30 to 32 years
  * 40 to 42 years

Exclusion Criteria:

* Non pregnant women
* Men
* No informed consent
* Age not included in inclusion criteria
* Major concomitant disease

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: three age groups
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Siegert, MD, DPharm, Phd, Principal Investigator — Technische Universität Dresden
Locations (1):
- Medizinische Fakultät der Technischen Universität Dresden, Dresden, Germany